CLINICAL TRIAL: NCT06308471
Title: The Effect of Baby Massage on Oral Motor Coordination Ability in Premature Babies
Brief Title: Effect of Baby Massage on Oral Motor Skills of Premature Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Nazire Arat, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ege üniversitesi
Record Dates: First submitted 2024-02-15; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Infant, Premature
Keywords: Oral feeding skills; Baby massage; Fucile protocol
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Baby massage was applied to the intervention group (20) of the study, and oral stimulation was applied with the Fucile protocol to the control group (20).
Who Masked: Participant, Outcomes Assessor
Masking Description: Professional nurses who evaluate nutrition do not know which group they belong to in the study.
  They do not know which group the premature babies are in due to their age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of baby massage (Experimental): Being between 28-33 weeks of gestation, Not having a congenital disease, Meeting the readiness criteria for oral feeding, Must be in the weight range of 1000-2000 grams
  Interventions: Other: Baby massage was applied to the intervention group (n=20) of the study
- Group of oral stimulation (Fucile Protocol) (Experimental): Being between 28-33 weeks of gestation, Not having a congenital disease, Meeting the readiness criteria for oral feeding, Must be in the weight range of 1000-2000 grams
  Interventions: Other: Oral stimulation

INTERVENTIONS:
Other: Baby massage was applied to the intervention group (n=20) of the study — The application was applied for 15 minutes every day for ten days, and oral feeding trials were video recorded. Feeding videos were evaluated by expert neonatal nurses using The Oral Feeding Scale without knowing the application group of the babies.
  Arms: Group of baby massage
Other: Oral stimulation — The application was applied for 15 minutes every day for ten days, and oral feeding trials were video recorded. Feeding videos were evaluated by expert neonatal nurses using The Oral Feeding Scale without knowing the application group of the babies.
  Arms: Group of oral stimulation (Fucile Protocol)

SUMMARY:
This experimental research was conducted in a single-blind, block randomized controlled design type.

The primary purpose of the study is to examine the effect of premature baby massage on oral motor coordination skills. The secondary aim is to evaluate the consistency of use of The Oral Feeding clinical scale in premature babies in Turkey.

As a result of the power analysis, baby massage was applied to the intervention group (n = 20) and oral stimulation with the Fucile protocol was applied to the control group (n = 20).

Comparative results were evaluated statistically.

DETAILED DESCRIPTION:
The Effect of Baby Massage on Oral Motor Coordination Ability in Prematures Purpose: The primary purpose of the study is to examine the effect of premature baby massage on oral motor coordination skills. The secondary aim is to evaluate the consistency of use of The Oral Feeding clinical scale in premature babies in Turkey.

Method: The research was a single-blind, block randomized controlled design type and data was collected between September 2021 and May 2023. Baby massage was applied to the intervention group (n=20) of the study, and oral stimulation was applied with the Fucile protocol to the control group (n=20). The applications were applied for 15 minutes every day for ten days, and oral feeding trials were video recorded. Feeding videos were evaluated by expert neonatal nurses using The Oral Feeding Scale. Descriptive statistical methods, Fisher test, chi-square analysis, dependent and independent t test, Mann Whitney U test, one-way analysis of variance, Kruskal Wallis test, Pearson and Spearman correlations were used to evaluate the research results.

ELIGIBILITY:
Inclusion Criteria:

* Being between 28-33 weeks of gestation,
* Not having a congenital disease,
* Clinical findings are stable and normal,
* It meets the readiness criteria for oral feeding,
* Being fed at full dose via Oral/Nasogastric tube and having never attempted oral intake before,
* It must weigh between 1000-2000 grams
* Parents give their consent to participate in the research and record video.

Exclusion Criteria:

* Premature babies of parents who did not give consent to participate in the study,
* Premature babies of parents who gave up participating in the study at any stage of the study,
* Physiological stability was impaired during the data collection process; Premature babies who require oxygen support and/or mechanical respirators,
* Conditions that disrupt clinical stability such as intracranial bleeding, necrotizing enterocolitis, neonatal sepsis are included in the process.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
time for first oral feeding | up to 36th week of gestation
  assessment of feeding skills
time for full oral feeding | up to 38th week of gestation
  assessment of feeding skills

SECONDARY OUTCOMES:
discharge time | up to 40th week of gestation
  time to hospital discharge (related to feeding ability)

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I want to think about sharing